CLINICAL TRIAL: NCT05039411
Title: A Phase I Study of the Safety of Allogeneic Human Umbilical Cord Mesenchymal Stem Cells (UC-MSCs) for Perianal Fistulas in Patients With Crohn's Disease
Brief Title: Safety of Allogeneic Human Umbilical Cord Mesenchymal Stem Cells (UC-MSCs) to Treat Perianal Fistulas w/ Crohn's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CryoCord Sdn Bhd (Industry)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCSB-CT-PF-01-2021 (Ver4.0)
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Perianal Fistula Due to Crohn's Disease; Fistula in Ano
Keywords: Perianal fistula; Crohn's Disease; Umbilical cord mesenchymal stem cells (UC-MSCs); Allogeneic stem cells
MeSH Terms: conditions — Rectal Fistula; Crohn Disease

STUDY DESIGN:
Intervention Model Description: All patients will receive a total of 60 million cells per visit for 5 consecutive visits, with a 6-12 weeks interval between the injections. If the patient is completely healed during any course of stem cell injections, subsequent stem cell treatments can be discontinued. However, patients will still be required to undergo regular follow-up examinations, including physical examinations and other medical tests, until the study is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PF2020-CELL (UC-MSCs) - Allogeneic Human Umbilical Cord Mesenchymal Stem Cells (Experimental): A total of 60 million PF2020-CELL (UC-MSCs) will be injected locally around the fistula tract, with a separation of 1 cm between injections. All patients will receive a total of 60 million cells per visit for 5 visits, with a 6 - 12 weeks interval between the injections. If the patient is completely healed during any course of stem cell injections, subsequent stem cell treatments can be discontinued. However, patients will still be required to undergo regular follow-up examinations, including physical examinations and other medical tests, until the study is completed.
  Interventions: Biological: PF2020-CELL (UC-MSCs) - Allogeneic Human Umbilical Cord Mesenchymal Stem Cells

INTERVENTIONS:
Biological: PF2020-CELL (UC-MSCs) - Allogeneic Human Umbilical Cord Mesenchymal Stem Cells — All patients will receive a total of 60 million PF2020-CELL (UC-MSCs) cells per treatment visit.

SUMMARY:
Objectives:

Primary: To demonstrate the safety of allogeneic UC-MSCs administered by injection for complex perianal fistulas in patients with Crohn's disease

Secondary: To determine the efficacy of a single/multiple allogeneic UC-MSCs injection in improving complex perianal fistula complications and (re-epithelialization of the external openings).

DETAILED DESCRIPTION:
Design and Investigation:

Number of Patients: 5 (including a consideration of 20% [1 patient] dropout from the trial)

Dosage and mode of administration Dosage: A total of 60 million PF2020-CELL (UC-MSCs) will be injected locally around the fistula tract, with a separation of 1 cm between injections. All patients will receive a total of 60 million cells per visit for 5 visits, with a 6 - 12 weeks interval between the injections. If the patient is completely healed during any course of stem cell injections, subsequent stem cell treatments can be discontinued. However, patients will still be required to undergo regular follow-up examinations, including physical examinations and other medical tests, until the study is completed.

Mode of administration: The procedure involves localizing the fistulous tract, performing curettage and closing the internal opening, and the injection of PF2020-CELL (UC-MSCs). The indicated dose of PF2020-CELL (UC-MSCs) will be injected starting from the tissues around the internal orifice or orifices and then progressing towards the external opening.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women age 18 years and above.
* Diagnosis of perianal fistulae associated with Crohn's disease refractory to medical therapy.
* Presence of perianal fistula(s) with a maximum of 2 internal openings and a maximum of 3 external openings based on clinical assessment.
* Fit for surgery.

Exclusion Criteria:

* Informed consent refusal.
* Pregnancy or breastfeeding women.
* Current diagnosis of active cancer or remission for less than 5 years.
* Evidence of active sepsis or significant localised infection.
* Patients with HIV, HBV, HCV or treponema infection, whether active or latent.
* Patients with documented allergies.
* Patients who have received infliximab or any other biologics in the 4 weeks before the cell treatment administration.
* Patients currently receiving, or having received within 1 month prior to enrollment into this clinical trial, any investigational drug.
* Patients with any other co-morbidity/ co-pathologies which is deemed as contraindication to stem cells infusion (infection, administration of steroids).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
No incidence of treatment-emergent adverse events (TEAEs) | Throughout study completion, an average of 1.5 year
  example of TEAEs are pyrexia (non-persistent fever, <38.5°C), infection, perianal abscess, enlargement of fistula & allergic reaction.

SECONDARY OUTCOMES:
Clinical healing | Visits 5, 9, 13, 17, 21 (approximately 6 to 12 weeks between visits)
  Mainly on re-epithelialization of external opening

CONTACTS AND LOCATIONS:
Overall Officials: April Camilla Roslani, Prof. Dr., Principal Investigator — Department of Surgery, Faculty of Medicine, University of Malaya
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No